CLINICAL TRIAL: NCT02617576
Title: Flavoring Oral Contrast for MR Enterography
Status: Withdrawn | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1507M76622
Record Dates: First submitted 2015-11-16; First posted 2015-12-01 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Taste, Altered
MeSH Terms: conditions — Dysgeusia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Flavored contrast: This group of patients will have the choice to flavor their contrast.
- Unflavored contrast: This group of patients will drink the contrast without flavoring.

SUMMARY:
To determine if patient satisfaction, participation, and image quality improves with flavored oral contrast for MR enterography.

DETAILED DESCRIPTION:
Volumen is an oral contrast agent used in MR imaging of the bowel. It has an unpleasant taste which makes it difficult for pediatric patients, especially sick pediatric patients, to drink. There are other contrast materials used in the department that are flavored to improved patient participation. The investigators hope to determine a way to flavor Volumen to improve patient participation. In doing so, the investigators hope to also improve patient satisfaction as well as imaging quality.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients having a MR enterography

Exclusion Criteria:

* sedated patients

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric patients undergoing MR enterography examinations
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
the number of patients that prefer flavored contrast | one year
  the number of patients that prefer flavored contrast will be evaluated by a questionaire
bowel diameter measurements on MR Enterography | one year
  bowel diameter measurements will be made by two radiologists on MR Enterography

CONTACTS AND LOCATIONS:
Overall Officials: Kelly Dietz, MD, Principal Investigator — University of Minnesota